CLINICAL TRIAL: NCT02252120
Title: Laryngeal Mask Airway Supreme Versus Laryngeal Tube in Non-paralysed, Anesthetized Children. A Randomized, Crossover Study Assessing Oropharyngeal Leak Pressure and Fiberoptic Position Using the Size 2
Brief Title: Laryngeal Mask Airway Supreme Versus Laryngeal Tube
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Schulthess Klinik (Other)
Collaborators: University of Salzburg (Other)
Responsible Party: Principal Investigator, ChristianKeller, PD Dr. med. M.Sc., Schulthess Klinik
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Schulthess_Anä_4
Record Dates: First submitted 2014-09-17; First posted 2014-09-29 (Estimated); Last update posted 2014-09-29 (Estimated); Status verified 2014-09

CONDITIONS: Adverse Anesthesia Outcome

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Supreme (Active Comparator): Supreme LMA
  Interventions: Device: Supreme; Device: Laryngeal Tube
- Laryngeal Tube (Active Comparator): Laryngeal tube LTSII
  Interventions: Device: Supreme; Device: Laryngeal Tube

INTERVENTIONS:
Device: Supreme
Device: Laryngeal Tube

SUMMARY:
The investigators test the hypothesis that oropharyngeal leak pressure and fiberoptic position differ between the size 2 LMA SupremeTM and the Laryngeal Tube LTS IITM in non-paralyzed anaesthetized pediatric patients

DETAILED DESCRIPTION:
The Laryngeal Tube LTS IITM (VBM-Medizintechnik GmbH, Sulz a.N, Germany) is a well established reusable latex free, extraglottic airway device. A proximal (pharyngeal) and a distal (esophageal) cuff are inflated with a single cuff pilot line. In between lies the ventilation orifice. The LMA SupremeTM (Teleflex San Diego, CA, USA) is a single use well studied laryngeal mask airway. Both devices have a drain tube to allow access to the gastrointestinal tract. Actually there are no studies comparing Laryngeal Tube LTS IITM and LMA SupremeTM use in small children. Therefore the aim of this study was to evaluate the clinical performance of the Laryngeal Tube LTS IITM compared to the LMA SupremeTM. The investigators hypothesized that design differences should lead to differences in efficacy of seal and anatomic position. In this randomized, crossover study, the investigators test the hypothesis that in non-paralyzed pediatric patients the oropharyngeal leak pressure and fiberoptic position differs between the size 2 Laryngeal Tube LTS IITM and the LMA SupremeTM.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II
* age 1.5 - 9 years
* minor surgery
* extraglottic airway device

Exclusion Criteria:

* age (<18 months, >9 years)
* weight (<10 kg, >25 kg)
* a known difficult airway
* risk of aspiration

Ages: 18 Months to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2014-01; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Oropharyngeal leak pressure | 5 Min
  Oropharyngeal leak pressure was determined by closing the expiratory valve of the anaesthesia breathing system and a fixed gas flow of 3 l minute-1. The airway pressure at which an equilibrium was reached was noted (maximum allowed 40 cm H2O).

SECONDARY OUTCOMES:
Fiberoptic position | 5 Min
  The airway tube view was scored using an established scoring system (4=only vocal cords visible; 3=vocal cords plus posterior epiglottis; 2=vocal cords plus anterior epiglottis; 1=vocal cords not seen)

OTHER OUTCOMES:
Ease of insertion | 1 Min
  We allowed one attempt before considering a failure, defining failed insertion by any of the following criteria:
  1) failed passage into the pharynx; 2) malposition (air leaks); and 3) ineffective ventilation (maximum expired tidal volume <4 ml kg-1 or end-tidal CO2 > 50 mm Hg (if correctly positioned). ). Insertion time was defined as the interval between picking up the prepared device and successfully placement. After placement effective ventilation was tested by observation of chest wall movement and capnometric curve trace. If insertion failed the etiology was signed on the CRF. After a first insertion attempt one single attempt with the guiding technique was allowed.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Keller, MD, M.Sc., Principal Investigator — Schulthess Klinik, Lengghalde 2, 8008 Zürich